CLINICAL TRIAL: NCT01105039
Title: Early Pain Pattern and Its Components After Laparoscopic Inguinal Hernia Repair
Brief Title: Detailed Pain Pattern After Laparoscopic Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Mette Astrup Tolver/MD., ph.d.-student, University Hospital Koge, gastroabdominal department
Other Study IDs: SJ-125X
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-02

CONDITIONS: Inguinal Hernia; Femoral Hernia
Keywords: Pain pattern; overall pain; incisional pain; shoulder pain; visceral pain
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Shoulder Pain; Visceral Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lap. hernia repair: undergoing laparoscopic groin hernia repair

SUMMARY:
Pain after laparoscopic groin hernia repair consist of different pain components (overall pain, shoulder pain, incisional pain and visceral pain). Thus it is important to find out which of these pain components that is most severe, so intervention can be targeted.

DETAILED DESCRIPTION:
Details about the components of early pain after laparoscopic groin hernia repair are lacking. A description of each component (overall pain, shoulder pain,incisional pain and visceral pain) is needed, so intervention against the different pain components can be targeted.

Patients fill out questionnaires about pain before operation and day 0-3 after operation.

ELIGIBILITY:
Inclusion Criteria:

* men
* 18-69 years
* uni- or bilateral hernia
* ASA I-II
* Danish speaking

Exclusion Criteria:

* bad compliance
* acute operation
* daily intake of opioids

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are consecutively included in this study. They are all undergoing elective laparoscopic groin hernia repair.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Overall pain during coughing (visual analog scale) | 3 days

SECONDARY OUTCOMES:
shoulder pain during coughing (visual analog scale and verbal rating scale) | 3 days
incisional pain during coughing (visual analog scale and verbal rating scale) | 3 days
visceral pain during coughing (visual analog scale and verbal rating scale) | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Mette A Tolver, M.D., Principal Investigator — Koge Hospital
Locations (1):
- University Hospital Koge, Køge, Sealand, Denmark